CLINICAL TRIAL: NCT05809843
Title: Deep Learning in Vascular and Structural Retinal Changes in Diabetic Patients Undergoing Artificial Pancreas Device
Brief Title: OCT and OCT-A Deep Learning in Diabetic Patients Wiht Artificial Pancreas Device
Status: Completed | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Ciro Costagliola, professor, Federico II University
Other Study IDs: 2403/2023
Record Dates: First submitted 2023-03-27; First posted 2023-04-12 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Type 1 Diabetes Mellitus With Artificial Pancreas Device

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- rype 1 diabetc patients with artificial pancreas device
  Interventions: Device: hybrid artificial pancreas systems (CSII)
- healthy patients matched age and sex without diabetes and ocular disease

INTERVENTIONS:
Device: hybrid artificial pancreas systems (CSII) — artificial device that adjust the patient's glycemic levels with insulin doses appropriate to the patient's blood glucose
  Groups: rype 1 diabetc patients with artificial pancreas device

SUMMARY:
This study evaluates the ability of deep learning to improve the knowledge about structural and vascular retinal changes in diabetic patients undergoing artificial pancreas device, using optical coherence tomography angiography.

DETAILED DESCRIPTION:
hybrid artificial pancreas systems (CSII) are able to adjust the type 1 diabetic patient's glycemic levels with insulin doses appropriate to the patient's blood glucose.

The optical coherence tomography angiography represents a novel and noninvasive diagnostic technique that allows a detailed and quantitative analysis of retinal and choriocapillary vascular features.

The study evaluates the changes in optical coherence tomography angiography features in diabetic patients undergoing artificial pancreas device, elaborating these data with artificial intelligence.

ELIGIBILITY:
Inclusion Criteria:

* • age older than 18 years

  * diagnosis of type 1 diabetes
  * treatment with artificial pancreas device
  * absence of previous ocular surgery and congenital eye diseases.
  * absence of errors of refraction
  * absence of lens opacities
  * absence of low-quality OCT and OCTA images

Exclusion Criteria:

* age younger than 18 years
* previous ocular surgery and congenital eye diseases
* errors of refraction
* lens opacities
* low-quality OCT and OCTA images

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The participans were older than 18 years with diagnosis of type 1 diabetes treated with artificial pancreas device. They did not present other ophthalmological disease
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2023-01-30 (Actual); Primary Completion 2023-03-23 (Actual); Study Completion 2023-03-23 (Actual)

PRIMARY OUTCOMES:
The measurements of retinal and choriocapillary vessel density in type 1 diabetic patients undergoing artificial pancreas device | up to 3months
  The parameters analyzed by optical coherence tomography angiography were: retinal and choriocapillary vessel density matched with clinical parameters resulted from the artificial pancreas device

CONTACTS AND LOCATIONS:
Locations (1):
- University of Naples "Federico II", Naples, Italy